CLINICAL TRIAL: NCT03434717
Title: Optimized Rehabilitation Following Primary Breast Cancer Surgery - Systematic Screening as a Tool for Individualised Rehabilitation: Study Protocol for the RE-SCREEN Randomized Controlled Trial
Brief Title: Optimized Rehabilitation Following Primary Breast Cancer Surgery
Acronym: RE-SCREEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RESCREEN
Record Dates: First submitted 2018-01-15; First posted 2018-02-15 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Rehabilitation; Breast Neoplasms; Psychological Distress
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (high distress) (Experimental): Control group receiving care as usual
  Interventions: Other: Care as usual
- Individualised rehabilitation (Experimental): Patients with high distress receive the intervention "individualized rehabilitation" including evaluation of individual needs and based on that physical, psychological or social interventions to promote rehabilitation.
  Interventions: Other: Individualised rehabilitation
- Control group (low distress) (Experimental): Control group receiving care as usual
  Interventions: Other: Care as usual

INTERVENTIONS:
Other: Individualised rehabilitation — Patients will get access/support to individualised rehabilitation based on their needs identified through the distress thermometer
  Arms: Individualised rehabilitation
Other: Care as usual — Patients will get care as usual
  Arms: Control (high distress); Control group (low distress)

SUMMARY:
This study aims to evaluate the effects of an intervention based on systematic screening of psychological distress as the basis for individualised support and rehabilitation following primary breast cancer surgery focusing on psychological , physical and health-economics outcomes. The aim is also to illuminate patients' and relatives' experiences and need of support during the rehabilitation .

DETAILED DESCRIPTION:
Breast cancer survivors are known to suffer from remaining problems from their treatment after surgery. Despite numerous of studies evaluating the effect of various rehabilitation programs it is know that patients often receive rehabilitation recommendations that are general rather than individualised to their needs. The large amount of studies within this area have contributed to knowledge about potential beneficial rehabilitation interventions for these patients but there is still a lack of knowledge about how patients specific needs of rehabilitation can be identified and how health care can adjust and individualize rehabilitation to optimize rehabilitation. This study aims to evaluate the effects of an intervention based on systematic screening of psychological distress as the basis for individualised support and rehabilitation following primary breast cancer surgery focusing on psychological , physical and health-economics outcomes. The aim is also to illuminate patients' and relatives' experiences and need of support during the rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Undergone treatment for primary breast cancer
* ≤18 years old
* Ability to communicate in Swedish
* Written informed consent

Exclusion Criteria:

* Recurrent disease
* Palliative diagnosis
* Pregnancy
* Prior history of breast cancer
* Inability to participate in the study due to cognitive impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 643 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Psychological Distress | Instrument will be answered approximately 1 week pre-operative and after surgery at 2 weeks, 3 ,6 ,9 and 1, 2 and 3 years postoperative. Evaluating change over time.
  Psychological Distress measured by the "Distress thermometer". A instrument that the patients answer themselves measuring the level of distress and the potential problems the may have.

SECONDARY OUTCOMES:
General Quality of life | Instrument will be answered approximately 1 week pre-operative and after surgery at 2 weeks, 3 ,6 ,9 and 1, 2 and 3 years postoperative. Evaluating change over time.
  The instrument QLQ-C30 is developed by the EORTC (European Organization for Research and Treatment of Cancer) and measurers quality of life
Information needs | Instrument will be answered approximately 1 week pre-operative and after surgery at 2 weeks, 3 ,6 ,9 and 1, 2 and 3 years postoperative. Evaluating change over time.
  The INFO35 instrument is developed by the EORTC and measures the patients perception of information received
Resilience | Instrument will be answered approximately 1 week pre-operative and after surgery at 2 weeks, 3 ,6 ,9 and 1, 2 and 3 years postoperative. Evaluating change over time.
  Conner-Davidsson Resilience scale (CD-RISC) will be used to measure patients resilience trough 25 questions ranging from 0-4. Lower scores indicates more problems
Life style changes | Instrument will be answered approximately 1 week pre-operative and after surgery at 2 weeks, 3 ,6 ,9 and 1, 2 and 3 years postoperative. Evaluating change over time.
  Life style changes will be measured by single items concerning exercise (amount hours of physical activity/day), Body mass index (based on weight and length), alcohol (units/glasses/ day) and tobacco habits (yes/no)
Health economics | Evaluations will be conducted after data collection is finished. 6 months and one year after inclusion.
  Cost-effectiveness analysis will be performed by evaluations of health care consumption (number of and total cost of health care visits) and by evaluating sickness absence (number of days)
Breast cancer specific quality of life | Instrument will be answered approximately 1 week pre-operative and after surgery at 2 weeks, 3 ,6 ,9 and 1, 2 and 3 years postoperative. Evaluating change over time.
  The instrument QLQ-BR23 is developed by the EORTC (European Organization for Research and Treatment of Cancer) and measurers diagnose specific quality of life
Satisfaction with care | Instrument will be answered approximately 1 week pre-operative and after surgery at 2 weeks, 3 ,6 ,9 and 1, 2 and 3 years postoperative. Evaluating change over time.
  Singel items focusing on satisfaction with care

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Malmström, PhD, Principal Investigator — Lund university, department of health siences, Lund
Locations (1):
- Skåne university hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olsson IM, Dykes C, Ryden L, Olsson-Moller U, Malmstrom M. Experiences of rehabilitation one year after breast cancer diagnosis-A focus group study from the ReScreen randomized controlled trial. PLoS One. 2025 Feb 13;20(2):e0315814. doi: 10.1371/journal.pone.0315814. eCollection 2025. PMID 39946344
- [Derived] Malmstrom M, Holst-Hansson A, Olsson Moller U. The complexity of needs and roles of family members during breast cancer rehabilitation: a qualitative study. BMC Cancer. 2024 Nov 21;24(1):1430. doi: 10.1186/s12885-024-13200-x. PMID 39567939
- [Derived] Olsson Moller U, Ryden L, Malmstrom M. Systematic screening as a tool for individualized rehabilitation following primary breast cancer treatment: study protocol for the ReScreen randomized controlled trial. BMC Cancer. 2020 May 29;20(1):484. doi: 10.1186/s12885-020-06815-3. PMID 32471390